CLINICAL TRIAL: NCT00275444
Title: Double-blind, Randomized, Dose Optimization Trial of Three Doses of Tipranavir Boosted With Low Dose Ritonavir (TPV/RTV) in Multiple Antiretroviral Drug-experienced Subjects
Brief Title: 3 TPV/RTV Doses in Multiple ARV Experienced Patients - Tipranavir Dose Defining Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1182.52
Record Dates: First submitted 2006-01-09; First posted 2006-01-12 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir

INTERVENTIONS:
Drug: Tipranavir

SUMMARY:
A dose defining study of the protease inhibitor tipranavir (TPV), boosted with low dose ritonavir (RTV). Three dose combinations of TPV/RTV are administered to multiple antiretroviral experienced patients and the dose that achieves the best efficacy and safety as determined by evaluation of 2, 8, and 24-week virologic response and adverse event and laboratory profile measures would be selected for further clinical study.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent prior to trial participation.
* Human immunodeficiency virus 1 (HIV-1) infected males or females > 18 years of age.
* At least 3 months experience taking Nucleoside reverse transcriptase inhibitors (NRTIs), Non-nucleoside reverse transcriptase inhibitor (NNRTIs), and Protease inhibitors (PIs).
* Current PI-based Antiretroviral (ARV) medication regimen for at least 3 months prior to randomization, and at least 3 months experience taking at least one other PI-based regimen.
* HIV-1 viral load ≥1000 copies/mL at screening.
* Genotypic resistance report indicating one or more primary PI resistance mutation(s), including 30N, 46I/L, 48V, 50V, 82A/F/T, 84V or 90M.
* Availability of 2 or more non-PI ARV medications by genotypic resistance testing, i.e. 2 drugs tested as "no evidence of resistance" or "possible resistance".
* Acceptable screening laboratory values that indicate adequate baseline organ function.
* Laboratory values are considered to be acceptable if severity is no higher than Grade 3 Gamma glutamyl transferase (GGT), Grade 2 cholesterol or triglycerides, and no higher than Grade 1 for all other tests based on the "Division of Acquired Immune Deficiency Syndrome" of National Institute of Health, USA - DAIDS - Grading Scale. All laboratory values outside these limits are subject to approval by Boehringer Ingelheim (BI).
* Further inclusion criteria apply.

Exclusion criteria:

* ARV medication naïve.
* Only one or no available ARV medications as determined by genotypic resistance testing.
* Female subjects who:

  * have a positive serum pregnancy test at screening or during the study;
  * are breast feeding;
  * are planning to become pregnant;
  * are not willing to use two methods of contraception to include at least one barrier method (e.g. latex condom plus spermicidal jelly/foam).
* Any active opportunistic infection within 60 days before study entry.
* Active Hepatitis B (HCB) or Hepatitis C (HCV) disease defined as HBsAg positive or HCV RNA positive with Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) > Grade 1.
* Prior tipranavir use.
* Use of investigational medications within 30 days before study entry or during the trial.Some expanded access drugs may be acceptable; must be approved by BI. Tenofovir, investigational at time of preparation of this protocol, is acceptable.
* Use of concomitant drugs which may significantly reduce plasma levels of the study medications.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2002-03-29 (Actual); Primary Completion 2003-01-20 (Actual)

PRIMARY OUTCOMES:
Virologic response after 2 weeks of functional monotherapy | At week 2

SECONDARY OUTCOMES:
Virologic response after 8 and 24 weeks of therapy and adverse event and laboratory safety measures. | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (62):
- United States (38):
  - Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - Living Hope Clinical Trials, Inc., Long Beach, California
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Vincent Lombardi Cancer Center, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - 1501 N.W. 9th Ave, Miami, Florida
  - Boehringer Ingelheim Investigational Site, Orlando, Florida
  - Boehringer Ingelheim Investigational Site, South Miami, Florida
  - Hillsborough County Health Dept., Tampa, Florida
  - Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - CORE Center, Chicago, Illinois
  - Rush-Presbytarian-St Luke's Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - HIV Outpatient Program (H.O.P), New Orleans, Louisiana
  - John's Hopkins University, Baltimore, Maryland
  - Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - Community Research Initiative of New England, Springfield, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - ID Care, Hillsborough, New Jersey
  - Boehringer Ingelheim Investigational Site, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - University of New York at Stony Brook, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, Annandale, Virginia
- Australia (2):
  - Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
- Canada (3):
  - Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Chest Institute - McGill University Health Centre, Montreal, Quebec
- France (6):
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de Chauliac, Montpellier
  - Hôpital Hôtel Dieu, Nantes
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital de la pitié Salpetrière, Paris
  - Hôpital Saint Louis, Paris
- Germany (4):
  - Epimed GmbH, Berlin
  - Klinik I für Innere Medizin der, Cologne
  - Klinikum der J.-W.-Goethe-Universität, Frankfurt am Main
  - Medizinische Poliklinik, München
- Italy (2):
  - Fondazione Centro S. Raffaele del Monte Tabor, Milan
  - IRCCS Policlinico San Matteo, Pavia
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Erasmus Medical Centre, Rotterdam
- Spain (4):
  - Hospital Clínico y Provincial de Barcelona - HIV, Barcelona
  - Boehringer Ingelheim Investigational Site, Madrid
  - Hospital La Paz., Madrid
  - Hospital Ramón y Cajal., Madrid
- 4th Floor Research Office (St Stephens Centre), London, United Kingdom